CLINICAL TRIAL: NCT01754779
Title: Pharmacological Therapy for Calcium Phosphate Urolithiasis
Brief Title: Treatment for Calcium Phosphate Kidney Stone Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Naim Maalouf, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 032012-058; R21DK097476-01 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-21 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Calcium Phosphate Kidney Stones
Keywords: calcium phosphate; urolithiasis; kidney stones; hypercalciuria
MeSH Terms: conditions — Urolithiasis; Kidney Calculi; Hypercalciuria | interventions — Citric Acid; Potassium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo, then Citric Acid, then Potassium Citrate (Experimental): Participants will receive at random, First intervention (1 week), then experience a washout period (1 week) and then receive Second Intervention (1 week) followed by another washout period of 1 week to finally receive the Third Intervention (1 week)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citric Acid; Dietary Supplement: Potassium Citrate
- Placebo, then Potassium Citrate, then Citric Acid (Experimental): Participants will receive at random, First intervention (1 week), then experience a washout period (1 week) and then receive Second Intervention (1 week) followed by another washout period of 1 week to finally receive the Third Intervention (1 week)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citric Acid; Dietary Supplement: Potassium Citrate
- Potassium Citrate, then Placebo, then Citric Acid (Experimental): Participants will receive at random, First intervention (1 week), then experience a washout period (1 week) and then receive Second Intervention (1 week) followed by another washout period of 1 week to finally receive the Third Intervention (1 week)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citric Acid; Dietary Supplement: Potassium Citrate
- Potassium Citrate, then Citric Acid, then Placebo (Experimental): Participants will receive at random, First intervention (1 week), then experience a washout period (1 week) and then receive Second Intervention (1 week) followed by another washout period of 1 week to finally receive the Third Intervention (1 week)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citric Acid; Dietary Supplement: Potassium Citrate
- Citric Acid, then Potassium Citrate, then Placebo (Experimental): Participants will receive at random, First intervention (1 week), then experience a washout period (1 week) and then receive Second Intervention (1 week) followed by another washout period of 1 week to finally receive the Third Intervention (1 week)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citric Acid; Dietary Supplement: Potassium Citrate
- Citric Acid, then Placebo, then Potassium Citrate (Experimental): Participants will receive at random, First intervention (1 week), then experience a washout period (1 week) and then receive Second Intervention (1 week) followed by another washout period of 1 week to finally receive the Third Intervention (1 week)
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Citric Acid; Dietary Supplement: Potassium Citrate

INTERVENTIONS:
Dietary Supplement: Placebo — 3 tablets twice daily of matching placebo during the placebo phase.
Dietary Supplement: Citric Acid — 3, 10 mEq tablets of H3Cit twice daily during the H3Cit phase (60 mEq H3Cit per day)
Dietary Supplement: Potassium Citrate — 2, 10 mEq K3Cit tablets and 1 placebo tablet twice daily during the K3Cit phase (40 mEq K3Cit per day)

SUMMARY:
The investigators will examine in two studies whether citric acid or potassium citrate can reduce calcium phosphate saturation in urine of Calcium Phosphate stone formers.

DETAILED DESCRIPTION:
We will examine in two short-term placebo-controlled cross-over metabolic studies whether citric acid or potassium citrate can reduce calcium phosphate saturation in urine of CaP stone formers.

The first study will be conducted in hypocitraturic CaP stone formers without hypercalciuria, and will compare the effects of potassium citrate, citric acid and placebo.

The second study will be conducted in hypercalciuric CaP stone formers on a thiazide diuretic who require potassium supplementation, and will compare the effects of potassium chloride alone, potassium chloride + citric acid, and potassium citrate alone. Physicochemical assays will be applied in addition to computer-based stone risk prediction programs to assess risk of stone recurrence.

ELIGIBILITY:
Inclusion Criteria:

Aim 1

* Hypocitraturic CaP stone formers
* urine citrate <320mg/d
* elevated pH as 24-hr urine pH above 6.40
* >21 years

Aim 2

* Hypercalciuric CaP stone formers
* 24hr urine calcium >250mg/d in women and >300mg/d in men prior to indapamide use
* high pH as >6.40 in the absence of urinary tract infection
* >21 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naim M Maalouf, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doizi S, Poindexter JR, Pearle MS, Blanco F, Moe OW, Sakhaee K, Maalouf NM. Impact of Potassium Citrate vs Citric Acid on Urinary Stone Risk in Calcium Phosphate Stone Formers. J Urol. 2018 Dec;200(6):1278-1284. doi: 10.1016/j.juro.2018.07.039. Epub 2018 Jul 20. PMID 30036516

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 41 patients who met inclusion criteria and were contacted for study enrollment, a total of 13 subjects agreed to enroll and were consented and each participant was evaluated during 3 phases in randomized order.
Period: First Intervention (1 Week)
Arm/Group | Placebo, Then Citric Acid, Then Potassium Citrate | Placebo, Then Potassium Citrate, Then Citric Acid | Potassium Citrate, Then Placebo, Then Citric Acid | Potassium Citrate, Then Citric Acid, Then Placebo | Citric Acid, Then Potassium Citrate, Then Placebo | Citric Acid, Then Placebo, Then Potassium Citrate
Started | 2 | 1 | 2 | 3 | 3 | 2
Completed | 2 | 1 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo, Then Citric Acid, Then Potassium Citrate | Placebo, Then Potassium Citrate, Then Citric Acid | Potassium Citrate, Then Placebo, Then Citric Acid | Potassium Citrate, Then Citric Acid, Then Placebo | Citric Acid, Then Potassium Citrate, Then Placebo | Citric Acid, Then Placebo, Then Potassium Citrate
Started | 2 | 1 | 2 | 3 | 3 | 2
Completed | 2 | 1 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Week)
Arm/Group | Placebo, Then Citric Acid, Then Potassium Citrate | Placebo, Then Potassium Citrate, Then Citric Acid | Potassium Citrate, Then Placebo, Then Citric Acid | Potassium Citrate, Then Citric Acid, Then Placebo | Citric Acid, Then Potassium Citrate, Then Placebo | Citric Acid, Then Placebo, Then Potassium Citrate
Started | 2 | 1 | 2 | 3 | 3 | 2
Completed | 2 | 1 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | Placebo, Then Citric Acid, Then Potassium Citrate | Placebo, Then Potassium Citrate, Then Citric Acid | Potassium Citrate, Then Placebo, Then Citric Acid | Potassium Citrate, Then Citric Acid, Then Placebo | Citric Acid, Then Potassium Citrate, Then Placebo | Citric Acid, Then Placebo, Then Potassium Citrate
Started | 2 | 1 | 2 | 3 | 3 | 2
Completed | 2 | 1 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Week)
Arm/Group | Placebo, Then Citric Acid, Then Potassium Citrate | Placebo, Then Potassium Citrate, Then Citric Acid | Potassium Citrate, Then Placebo, Then Citric Acid | Potassium Citrate, Then Citric Acid, Then Placebo | Citric Acid, Then Potassium Citrate, Then Placebo | Citric Acid, Then Placebo, Then Potassium Citrate
Started | 2 | 1 | 2 | 3 | 3 | 2
Completed | 2 | 1 | 2 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Citric Acid, Then Potassium Citrate | Placebo, Then Potassium Citrate, Then Citric Acid | Potassium Citrate, Then Placebo, Then Citric Acid | Potassium Citrate, Then Citric Acid, Then Placebo | Citric Acid, Then Potassium Citrate, Then Placebo | Citric Acid, Then Placebo, Then Potassium Citrate | Total
Number analyzed (Participants) | 2 | 1 | 2 | 3 | 3 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (9.2) | 34.8 | 49.2 (27.9) | 41.4 (24.5) | 45.6 (11.8) | 35.6 (1.3) | 41 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 2 | 3 | 2 | 11
  Male | 1 | 0 | 0 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 0 | 0 | 0 | 0 | 2 | 0 | 2
  White | 2 | 1 | 2 | 3 | 1 | 2 | 11
  Hispanic | 1 | 1 | 1 | 1 | 0 | 0 | 4
  Non-Hispanic | 0 | 0 | 1 | 2 | 3 | 2 | 8
Height [Mean (Standard Deviation); unit: metres] | 1.66 (0.13) | 1.58 | 1.56 (0.02) | 1.63 (0.18) | 1.69 (0.06) | 1.64 (0.05) | 1.63 (0.10)
Weight [Mean (Standard Deviation); unit: kg] | 74.2 (3.4) | 89.0 | 70.3 (18.0) | 56.7 (16.0) | 91.4 (11.0) | 53.8 (7.4) | 71.6 (18.5)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.9 (2.8) | 35.9 | 28.9 (8.0) | 21.2 (2.7) | 32.1 (2.1) | 20.2 (4.0) | 26.7 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Urinary Calcium Phosphate Saturation
Description: This variable represents a ratio of the calcium phosphate saturation in a given urine sample to the calcium phosphate saturation at the point of precipitation and hence this measure has no units.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: no units
Groups:
- Placebo: Placebo tablets twice daily
  Placebo: Matching placebo for both aims.
- Citric Acid: Citric acid tablets twice daily
  Citric Acid
- Potassium Citrate: Potassium Citrate tablets twice daily
  Potassium Citrate
Arm/Group | Placebo | Citric Acid | Potassium Citrate
Number analyzed (Participants) | 13 | 13 | 13
no units | 2.38 (1.07) | 1.97 (0.75) | 2.19 (0.96)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Placebo | Citric Acid | Potassium Citrate
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/13

LIMITATIONS AND CAVEATS:
The second study (in hypercalciuric Cap stone formers) was never conducted due to difficulties in recruitment and limited budget.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT01754779/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/79/NCT01754779/ICF_001.pdf